CLINICAL TRIAL: NCT03675334
Title: Clinical Comparison Between the Use of a Connective Tissue Graft or a Porcine Collagen Matrix (Mucoderm) for Treatment of Gingival Recessions Type 1: a Randomized Controlled Clinical Study.
Brief Title: Mucoderm or Connective Tissue Graft for Treatment of Gingival Recessions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, Phd, Ms, DDs. Chairman of Periodontolgy, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 58534216.5.0000.5419
Record Dates: First submitted 2018-09-10; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Gingival Recession
Keywords: clinical trial; root coverage; biomaterials; collagen matrix; coronally advanced flap
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Split-mouth clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The clinical parameters were screened by one single examiner that was not aware of the procedures
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Active Comparator): Active comparator: gingival recession
  the aim of this study is to compare if the collagen matrix graft is as efficient as a substitute for the connective graft used in root coverage of gingival recessions
  Interventions: Procedure: Root coverage with collagen matrix graft; Other: Basic periodontal treatment
- Control Group (Placebo Comparator): the aim of this study is to compare if the collagen matrix graft is as efficient as a substitute for the connective graft used in root coverage of gingival recessions. The control group was treated with the same technique as the collagen matrix graft.
  Interventions: Procedure: Root coverage with subepithelial connective tissue graft; Other: Basic periodontal treatment

INTERVENTIONS:
Procedure: Root coverage with collagen matrix graft — at one side, the root coverage have been done with a extended flap technique and collagen matrix graft. At the other side, the same technique was performed with connective graft.
  Arms: Test Group
Procedure: Root coverage with subepithelial connective tissue graft — at one side, the root coverage have been done with a extended flap technique and collagen matrix graft. At the other side, the same technique was performed with connective graft.
  Arms: Control Group
Other: Basic periodontal treatment — profilaxis, coronary polishing and scaling and root planning

SUMMARY:
Coronally advanced flap plus connective tissue graft (CTG) is the gold standard therapy for root coverage. The bioabsorbable porcine collagen matrix (CM) has been widely used in periodontal and mucogingival surgery as a substitute for CTG and has achieved similar results. The CM has the advantage of no need of a second surgical area and availability overcoming the limitations of donor site in autograft.

The aim of this study is to investigate the use of Mucoderm® in root coverage procedures combined with extended coronally positioned flap (ECAF), test group (TG), in comparison to the connective tissue graft associated with the ECAF, control group (CG).

ELIGIBILITY:
Inclusion Criteria:

* CEJ without significant damage;
* localized bilateral RT1 gingival recession ≥3 mm in the same arch

Exclusion Criteria:

* previous periodontal surgical treatment on the involved sites;
* smokers
* pregnants or lactating
* compromised systemic health and contraindications for periodontal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Root coverage after 6 months | 6 months
  Root coverage is measured by the difference between the gingival recession height at 6 months and baseline

SECONDARY OUTCOMES:
Keratinized tissue gain after 6 months | 6months
  The difference between keratinized tissue width and depth at 6 months and at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry of Ribeirao Preto - University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suzuki KT, de Jesus Hernandez Martinez C, Suemi MI, Palioto DB, Messora MR, de Souza SLS, Novaes AB Jr, Chaves Furlaneto FA, Taba M Jr. Root coverage using coronally advanced flap with porcine-derived acellular dermal matrix or subepithelial connective tissue graft: a randomized controlled clinical trial. Clin Oral Investig. 2020 Nov;24(11):4077-4087. doi: 10.1007/s00784-020-03280-x. Epub 2020 May 7. PMID 32382931